CLINICAL TRIAL: NCT05503017
Title: An Investigation of a Brief Psycho-Social Computerized Intervention Targeting the Error-Related Negativity and Balance N1 in Anxious Children
Brief Title: Computerized Intervention Targeting the Error-Related Negativity and Balance N1 in Anxious Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Norman Schmidt, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00003181; 1F32MH129076-01A1 (NIH)
Record Dates: First submitted 2022-08-10; First posted 2022-08-16 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Anxiety Disorders; Generalized Anxiety Disorder; Social Anxiety Disorder; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social; Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Psycho-social, computerized intervention targeting error sensitivity
- Control Condition (Active Comparator)
  Interventions: Behavioral: Psycho-social, computerized intervention on healthy lifestyle choices

INTERVENTIONS:
Behavioral: Psycho-social, computerized intervention targeting error sensitivity — The computer-based intervention is designed to directly reduce the sensitivity to errors through cognitive behavioral techniques. The intervention takes approximately 45 minutes and includes interactive quizzes, information, and behavioral tasks relevant to making mistakes, implications of making errors, and ways to deal with making mistakes, among other topics relevant to increased error sensitivity. The intervention uses developmentally appropriate language and stories that young children can relate to and understand.
  Arms: Intervention
Behavioral: Psycho-social, computerized intervention on healthy lifestyle choices — The computer-based control condition will be in the same format and duration as the active intervention, but instead focuses on self-care topics and healthy lifestyle choices (e.g., eating healthy foods and getting a good night sleep), unrelated to error sensitivity.
  Arms: Control Condition

SUMMARY:
Anxiety disorders are the most common form of psychopathology, and frequently begin in childhood, resulting in lifelong impairment. Increased brain activity after making mistakes, as reflected by the error-related negativity (ERN), is observed in people with anxiety disorders, even before disorder onset. The ERN is therefore of great interest as a potentially modifiable risk factor for anxiety. However, methodological issues can make the ERN difficult to measure.

Increased brain activity in response to a balance disturbance, as reflected by the balance N1, resembles the ERN, but does not share its methodological issues. The investigators' preliminary data demonstrate that the balance N1 and the ERN are associated in amplitude in adults, suggesting they may depend on the same brain processes. The balance N1 has never been investigated in individuals with anxiety disorders, but it increases in amplitude within individuals under anxiety-inducing environmental contexts. Further, balance and anxiety are related in terms of brain anatomy, daily behavior, disorder presentation, and response to treatment.

The present investigation will measure the ERN and the balance N1 in children (ages 9-12) with anxiety disorders, and further, how these brain activity measures change in response to a brief, 45-minute, computerized psychosocial intervention that was developed to reduce reactivity to errors, and has been shown to reduce the ERN. The investigators will recruit approximately 80 children with anxiety disorders, half of whom will be randomly assigned to the active intervention condition. The other half will be assigned to an active control condition, consisting of a different 45-minute computerized presentation. Participants assigned to the control condition can access the computerized intervention after participation in the study.

The purpose of this investigation is to test the hypothesis that the balance N1 and the ERN will be reduced to a similar extent after the intervention, to demonstrate that these brain responses arise from shared brain processes. Transfer of the effect of the psycho-social intervention to the balance N1 would provide insight into prior work demonstrating that balance training can alleviate anxiety in young children, and well-documented benefits of psychotherapy to balance disorders. Collectively, these data may guide the development of multidisciplinary interventions for the prevention and treatment of anxiety disorders in children.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking child
* Must be able to stand for 15 minutes without assistance
* Anxiety disorder (generalized anxiety disorder, social anxiety disorder, and/or obsessive-compulsive disorder)

Exclusion Criteria:

* Depression or attention-deficit hyperactivity disorder
* Significant medical condition, developmental disorder, or physical disability affecting the ability to stand
* Severe psychopathology (e.g., bipolar disorder, psychosis, thought disorder, neurological disease, severe or extreme suicide risk)
* Head injuries (over the past three months) that resulted in a loss of consciousness
* Absence of an English-speaking primary caregiver that can accompany the child to the laboratory visit.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Change in ERN after intervention | 1 hour
  The change in magnitude of the error-related negativity between baseline and reassessment after the intervention
Change in balance N1 after intervention | 1 hour
  The change in magnitude of the error-related negativity between baseline and reassessment after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Norman B Schmidt, PhD, Principal Investigator — Florida State University
Locations (1):
- FSU Psychology Building, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and statistical analysis plan will be available as posted on clinicaltrials.gov upon posting of summary results information (i.e., within 1 year of study completion). Deidentified data dictionaries will also be made publicly available upon posting of summary results information. The data dictionaries (in the form of a spreadsheet) will include at least the following: age, sex, assignment to intervention or control condition, and baseline and reassessment amplitudes of both the ERN and the balance N1. The processed waveforms from which the ERN and balance N1 amplitudes are measured will also be made publicly available in a ".mat" file, viewable in MATLAB. Once these are posted, the associated access link will be updated here.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available upon posting of summary results information within 1 year of study completion.
Access Criteria: Publicly available